CLINICAL TRIAL: NCT07189143
Title: The Effect of Silver Fir Branch Extract on Liver and Kidney Function
Brief Title: Silver Fir Safety in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0120-642/2017/5
Record Dates: First submitted 2025-08-19; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Safety / Toxicology; Liver Function; Kidney Function; Dietary Supplement; Healthy Volunteers
Keywords: Abies alba; Silver fir extract; Dietary supplement; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Belinal® Group (Experimental): Participants received Belinal® (Abies alba branch extract) capsules at a total daily dose of 900 mg (4 × 225 mg) for 14 consecutive days. The supplement was taken orally in divided doses throughout the day.
  Interventions: Dietary Supplement: Belinal® (Abies alba branch extract)

INTERVENTIONS:
Dietary Supplement: Belinal® (Abies alba branch extract) — Belinal® capsules, 900 mg/day (4 × 225 mg), orally for 14 consecutive days.

SUMMARY:
This study evaluated the safety of Belinal®, a dietary supplement made from silver fir (Abies alba) branch extract, in healthy volunteers. Fifteen adults took 900 mg of Belinal® daily for 14 days. Blood tests were performed at several time points to measure liver and kidney function (enzymes and other biochemical markers).

DETAILED DESCRIPTION:
This was a prospective, open-label, single-arm interventional study conducted to assess the toxicological safety of Belinal®, a standardized water extract from silver fir (Abies alba) branches. Belinal® contains polyphenols, including lignans, flavonoids, and phenolic acids, which have demonstrated various pharmacological activities in previous studies.

The study enrolled 15 healthy volunteers (8 men, 7 women; age range 37-55 years). Participants received Belinal® capsules at a total daily dose of 900 mg (4 × 225 mg) for 14 consecutive days.

The study design included three consecutive two-week periods:

Wash-out period: to eliminate potential effects of prior supplement use. Comparative period: to assess natural variability in laboratory parameters without supplementation.

Test period: during which participants consumed Belinal® daily. Safety was evaluated by measuring liver and kidney biochemical parameters (AST, ALT, ALP, GGT, bilirubin, urea, creatinine, uric acid) at baseline, day 14, day 28, and day 42. Adverse events were monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* Age 37-55 years
* Both sexes (male and female)
* Willingness to comply with study protocol and attend all study visits
* Signed informed consent

Exclusion Criteria:

* Known acute or chronic illness
* Use of any medications other than occasional analgesics (none were used by participants)
* Use of dietary supplements prior to or during the study
* Known mental illness (e.g., depression, psychosis, severe alcoholism, drug abuse)
* Consumption of more than 2 alcohol units per day (20 g ethanol, equivalent to ~2 dl wine, 5 dl beer, or 0.3 dl brandy)
* Participation in other research studies concurrently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Change in serum AST | Baseline, Day 14, Day 28, and Day 42.
  Change in aspartate aminotransferase (AST) to evaluate potential hepatotoxic effects. Unit of Measure: U/L
Change in serum ALT | Baseline, Day 14, Day 28, Day 42.
  Change in alanine aminotransferase (ALT) to evaluate potential hepatotoxic effects. Unit of Measure: U/L
Change in serum ALP | Baseline, Day 14, Day 28, Day 42.
  Change in alkaline phosphatase (ALP) levels to evaluate potential hepatobiliary effects. Unit of Measure: U/L
Change in serum GGT | Baseline, Day 14, Day 28, Day 42.
  Change in gamma-glutamyl transferase (GGT) levels to evaluate potential hepatobiliary effects. Unit of Measure: U/L
Change in serum bilirubin | Baseline, Day 14, Day 28, Day 42.
  Change in total bilirubin as a marker of liver function. Unit of Measure: µmol/L
Change in serum urea | Baseline, Day 14, Day 28, Day 42.
  Change in blood urea levels as a marker of kidney function. Unit of Measure: mmol/L
Change in serum creatinine | Baseline, Day 14, Day 28, Day 42.
  Change in serum creatinine levels as a marker of kidney function. Unit of Measure: µmol/L
Change in serum uric acid | Baseline, Day 14, Day 28, Day 42.
  Change in uric acid levels as a marker of kidney function. Unit of Measure: µmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Belinal® information — https://belinal.eu